CLINICAL TRIAL: NCT05761730
Title: The Efficacy of Orally Administered Dexamethasone in the Management of Symptomatic Irreversible Pulpitis Without Performing Pulpotomy : : A Single-arm Open Clinical Trial
Brief Title: Oral Dexamethasone for the Management of Symptomatic Irreversible Pulpitis Without Performing Pulpotomy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: May Samaha (Other)
Responsible Party: Sponsor-Investigator, May Samaha, Director of the medical library- Saint Joseph University, Saint-Joseph University
Organization: Saint-Joseph University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USJ-2022-212
Record Dates: First submitted 2023-02-15; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Irreversible Pulpitis
Keywords: "irreversible pulpitis " "mandibular molars " "pain" "pulpotomy" "dexamethasone"
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: The participants will be allocated to two groups randomly the aim of this randomized clinical study is to assess the effect of dexamethasone on the reduction of pain in mandibular molars with irreversible pulpitis, without performing conventional pulpotomy ( intervention group ) in comparison to pain following pulpotomy ( control group )
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control group (No Intervention): Patients suffering from acute pain due to symptomatic irreversible pulpitis on a lower mandibular molar . Conventional emergency treatment is performed . Pulpotomy is performed after inferior alveolar nerve block injection ( IANB )
- Intervention Group (Experimental): Patients suffering from acute pain due to symptomatic irreversible pulpitis on a lower mandibular molar . Short course orally administered dexamethasone after inferior alveolar nerve block injection without performing conventional pulpotomy
  Interventions: Drug: Dexamethasone Oral

INTERVENTIONS:
Drug: Dexamethasone Oral — For a patient suffering from an irreversible pulpitis on a lower mandibular molar , 4mg of dexamethasone are administered at baseline , after inferior alveolar nerve block injection and 4mg are administered 8 hours after the first dose at office
  Arms: Intervention Group

SUMMARY:
The efficacy of short course orally administered dexamethasone on the reduction of pain before conventional pulpotomy has not yet been demonstrated.

Therefore, the aim of this randomized clinical study is to assess the effect of dexamethasone on the reduction of pain in mandibular molars with irreversible pulpitis, without performing conventional pulpotomy in comparison to pain following pulpotomy.

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy patients (Category: American Society of Anesthesiologists class 1) (ASA House of Delegates 2014) aged between 18 and 40 years with mandibular molars diagnosed with symptomatic irreversible pulpitis and a radiographically normal periapical region were included. Diagnosis was based on clinical and radiographic examination and pulp sensibility testing. Teeth were included if they responded long-term to cold test, the cold test was performed by injecting a syringe filled with cold water at the level of the suspicious tooth and the adjacent teeth. Teeth with deep occlusal decay, old restoration with underlying decay, recent restoration or crown were included. Patients that agreed to be contacted by phone after the emergency visit until pain relief, that were available to come back after the emergency visit for complete endodontic treatment and who had the ability to understand the informed consent form and pain recording scales used within this study were included.

Exclusion Criteria:

Teeth with acute or chronic apical abscess, pulp necrosis, septum syndrome and open apices were excluded. Medically compromised patients, pregnant and lactating women were excluded. Patients having history of allergy to local anesthetic solutions or any of the experimental drugs, on long-term medications that influenced pain threshold, analgesics, steroids and/or antibiotics in the recent past 24 h, were also excluded from the trial. Patients that suffered from a viral disease in evolution (Hepatitis, Herpes Zoster, Ocular Herpes), have or had a history of tuberculosis, hypertension, renal insufficiency, adrenocortical dysfunction, epilepsy, systemic fungal infections, GUILLAIN-BARRE syndrome, peptic ulcers and gastro intestinal disorders were excluded. Patients with Temporomandibular joint disorders were excluded. Patients suffering from mental disabilities were also excluded.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | The pain was measured 4 times : 1- at baseline in the office on a visual analog scale , 2-8 hours after the first dose of dexa on a visual analog scale , 3- 12 hours after the first dose of dexa on a visual analog scale , 4- 24 hours afterthe first dose
  To measure the change of the intensity of pain on a visual analog scale at different time periods before and after the administration of dexamethasone in the intervention group and to measure pain before and after pulpotomy in the control group at different time periods

CONTACTS AND LOCATIONS:
Overall Officials: L'emira Sara CHEHAB, Principal Investigator — saint joseph university of beirut
Locations (1):
- Saint Joseph University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pochapski MT, Santos FA, de Andrade ED, Sydney GB. Effect of pretreatment dexamethasone on postendodontic pain. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2009 Nov;108(5):790-5. doi: 10.1016/j.tripleo.2009.05.014. Epub 2009 Sep 12. PMID 19748294
- [Background] Mehrvarzfar P, Esnashari E, Salmanzadeh R, Fazlyab M, Fazlyab M. Effect of Dexamethasone Intraligamentary Injection on Post-Endodontic Pain in Patients with Symptomatic Irreversible Pulpitis: A Randomized Controlled Clinical Trial. Iran Endod J. 2016 Fall;11(4):261-266. doi: 10.22037/iej.2016.2. PMID 27790253
- [Background] Krasner P, Jackson E. Management of posttreatment endodontic pain with oral dexamethasone: a double-blind study. Oral Surg Oral Med Oral Pathol. 1986 Aug;62(2):187-90. doi: 10.1016/0030-4220(86)90044-7. PMID 3528979
- [Background] Bidar M, Mortazavi S, Forghani M, Akhlaghi S. Comparison of Effect of Oral Premedication with Ibuprofen or Dexamethasone on Anesthetic Efficacy of Inferior Alveolar Nerve Block in Patients with Irreversible Pulpitis: A Prospective, Randomized, Controlled, Double-blind Study. Bull Tokyo Dent Coll. 2017;58(4):231-236. doi: 10.2209/tdcpublication.2016-0050. PMID 29269717